CLINICAL TRIAL: NCT05312645
Title: Diclofenac Gel in the Treatment of Cervicogenic Headache: A Randomized, Double-Blind, Controlled Trial
Brief Title: Diclofenac Gel in the Treatment of Cervicogenic Headache
Acronym: DITCH
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No Subjects Enrolled
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5230175
Record Dates: First submitted 2022-03-28; First posted 2022-04-05 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Cervicogenic Headache
Keywords: Headache; Cervicogenic; Diclofenac
MeSH Terms: conditions — Post-Traumatic Headache; Headache | interventions — Diclofenac; Petrolatum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Diclofenac Gel (Experimental): Nursing staff will apply 2 grams of diclofenac 1% gel topically to the posterior cervical region of the subject four times daily for 14 days. A questionnaire consisting of a Numeric Assessment Scale (NAS) and Headache Impact Test (HIT-6) will be administered at baseline (day 1), day 7, and at the study conclusion (day 14). A complete metabolic panel will obtained on day 0 and on day 14.
  Interventions: Drug: Diclofenac 1% Topical
- Control (Placebo Comparator): Nursing staff will apply a petroleum gel based compound topically to the posterior cervical region of the subject four times daily for 14 days. A questionnaire consisting of a Numeric Assessment Scale (NAS) and Headache Impact Test (HIT-6) will be administered at baseline (day 1), day 7, and at the study conclusion (day 14). A complete metabolic panel will obtained on day 0 and on day 14.
  Interventions: Other: Petroleum Jelly

INTERVENTIONS:
Drug: Diclofenac 1% Topical — 2 grams topically four times daily for 2 weeks to posterior cervical spine
  Arms: Diclofenac Gel
Other: Petroleum Jelly — 2 grams topically four times daily for 2 weeks to posterior cervical spine
  Arms: Control

SUMMARY:
The intervention will consist of the nursing staff applying 2 grams of diclofenac 1% gel topically to the posterior cervical region four times daily. The control group will receive petroleum jelly topically to the posterior cervical region four times daily. Patients will receive a pre-intervention and post-intervention survey incorporating the Numeric Assessment Scale and Headache Impact Test-6.

ELIGIBILITY:
Inclusion criteria:

1. 18-90 Years old
2. Subject must be able to consent for themselves
3. Hospitalized at Loma Linda East Campus Rehabilitation Hospital
4. English or Spanish speaking
5. Complain of a headache, caused by a disorder of the cervical spine and/or it's component (i.e. bony, disc and/or soft tissue elements) usually but not invariably accompanied by neck pain (Avijgan et al, 2019)).

Exclusion criteria:

1. Primary headache secondary to intracranial pathology (i.e. tumors)

   a. While TBI and Stroke patients can suffer headaches as a sequalae of their intracranial pathologies, it is not always the case that their headache is primarily secondary to their pathology but due to other etiologies such as cervicogenic headache or myofascial pain syndrome. History and physical examination by the medical team will help aid in determining the headache's etiology.
2. Patients on dual antiplatelet therapy

   a. Aspirin 81mg daily or Clopidogrel (or antiplatelet monotherapy) is acceptable
3. History of cervical spine procedures

   a. Spinal cord injury patients with cervical neck injuries that have required operative repair will be excluded from the study.
4. Nerve blocks within past 4 weeks or steroid injections within past 6 months.
5. Patients with fibromyalgia
6. Pregnant women
7. Chronic pain on continuous opiate regimen (use of opioids on most days >90 days)
8. Discharged in less than 14 days from acute inpatient rehabilitation
9. Any contraindication use per diclofenac gel package insert:

   1. Known hypersensitivity to diclofenac or any other components of the drug product
   2. History of asthma, uriticaria, or other allergic-type reactions after taking aspirin or other NSAIDs.
   3. In the setting of coronary artery bypass graft (CABG) surgery.
10. Development of adverse reaction resulting in discontinuation of diclofenac gel

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-08-21 (Actual); Study Completion 2024-08-21 (Actual)

PRIMARY OUTCOMES:
Pain Severity | Change between baseline and day 14 of treatment.
  Measured with the Numeric Assessment Scale (0 least severe, 10 most severe). This is a composite measurement between pre-intervention baseline and 14 days post-treatment.
Activities of Daily Living Function Assessment | Change between baseline and day 14 of treatment.
  Measured with Headache Impact Test-6 (score less than 49 indicates little to no impact on daily life, 50-55 indicates some impact, 56-59 indicates substantial impact, greater than 60 indicates severe impact). This is a composite measurement of activities of daily living function between pre-intervention baseline and 14 days post-treatment. Activities of daily living include, but are not limited to, household work, grooming, and social activities.

CONTACTS AND LOCATIONS:
Overall Officials: Duc Tran, MD, PhD, Principal Investigator — Loma Linda University
Locations (1):
- Tom Vi and Zapara Rehabilitation Pavillion, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No